CLINICAL TRIAL: NCT06582381
Title: Evaluation of Biomarkers for Predicting Macronutrient Intake
Acronym: Microdialysis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Texas A&M University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Marielle PKJ Engelen, PhD, Professor, Texas A&M University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 91-Micro2; R01DK136414 (NIH)
Record Dates: First submitted 2024-08-30; First posted 2024-09-03 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Glucose Metabolism; Amino Acid Metabolism
Keywords: amino acid; glucose; metabolism; microdialysis; nutrition; stable isotope; macronutrient; biomarker

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Laboratory staff and data scientists will not know the meals received when analyzing samples and initial statistical modeling
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy male older adults (Experimental): Eight predefined, commercially available meal is administered in a randomized fashion. Two meals are consumed 6 hours apart on each study day. Meals are selected to represent a range of fat, protein, and carbohydrate content.
  Interventions: Other: Meal set A; Other: Meal set B; Other: Meal set C; Other: Meal set D
- Healthy female older adults (Experimental): Eight predefined, commercially available meal is administered in a randomized fashion. Two meals are consumed 6 hours apart on each study day. Meals are selected to represent a range of fat, protein, and carbohydrate content.
  Interventions: Other: Meal set A; Other: Meal set B; Other: Meal set C; Other: Meal set D

INTERVENTIONS:
Other: Meal set A — morning meal: low carbohydrate, low protein, low fat afternoon meal: high carbohydrate, high protein, high fat
Other: Meal set B — morning meal: low carbohydrate, high protien, low fat meal afternoon meal: high carbohydrate, low protein, high fat meal
Other: Meal set C — morning meal: low carbohydrate, low protien, low fat meal afternoon meal: high carbohydrate, high protein, low fat meal
Other: Meal set D — morning meal: high carbohydrate, low protien, low fat meal afternoon meal: low carbohydrate, high protein, high fat meal

SUMMARY:
The goal of this clinical trial is to establish the relationship between macronutrient food intake and the resulting blood and intersticial fluid (ISF )levels of small molecule markers, as well as, validate wearable optical readers and data fusion algorithms to accurately predict individual-specific macronutrient availability in real time.

The study involves 1 screening visit of approximately 2 hours and up to 4 study days of approximately 14 hours. Subjects will be asked to arrive in the fasted state on all study days. Fasting prior to screening is not required. On the screening visit, body weight, height, and body composition by Dual-energy X-ray absorptiometry (DXA) will be measured. In addition, habitual dietary intake, physical activity level (PASE), and quality of life (SGRQ-C) will be assessed.

DETAILED DESCRIPTION:
On each study day, body weight and height will be measured. An in-dwelling catheter will be inserted in a peripheral vein of the lower arm or hand to enable blood sampling. The arm will be put in a hot box to allow collecting arterialized venous blood samples. After taking a baseline blood sample, the predefined meal will be consumed within 10 min. Small arterialized venous blood samples (5 ml) will subsequently be drawn multiple times. Samples will be collected in predefined tubes, plasma/serum separated, aliquoted, and stored at -80 deg. Celsius for later assays and/or send to a local accredited laboratory for the concentrations of amino acids and other parameters (including amino acids, fatty acids, glucose, insulin).

In the opposite limb, a commercially available microdialysis catheter will be placed in the forearm following standard operating procedures developed by the European Academy of Allergy & Clinical Immunology Task Force on Skin Microdialysis. Dialysate will be collected in 30-minute aliquots in microvials for the duration of the study day. Microvials will be weighed before and after sample collection. A syringe filled with perfusate containing mixture of stable tracer-labelled amino acids and glucose will be infused through the syringe pump at a controlled rate.

On each of the study days, subjects will consume two meals with defined composition of macronutrients eight hours apart.

ELIGIBILITY:
Inclusion criteria

* Ability to walk, sit down and stand up independently
* Age 50-75 years old
* Ability to lie in supine or slightly elevated position for approximately 13 hours
* BMI between 25 and 35
* Willingness and ability to comply with the protocol

Exclusion Criteria

* Established diagnosis of malignancy
* Established diagnosis of Insulin or non-Insulin Dependent Diabetes Mellitus
* History of untreated metabolic diseases including hepatic or renal disorder
* Currently on anticoagulants (i.e., warfarin, factor X inhibitors or direct thrombin inhibitors)
* History of deep vein thrombosis, pulmonary embolisms, or known clotting disorders
* Presence of acute illness or metabolically unstable chronic illness
* Recent myocardial infarction (less than 1 year)
* Known allergy or intolerance to any of the meal components
* Any other condition according to the PI or nurse that was found during the screening visit, that would interfere with the study or safety of the patient
* Failure to give informed consent or Investigator's uncertainty about the willingness or ability of the participant to comply with the protocol requirements

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2023-12-06 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Glucose metabolism | Up to 14 hours per study visit, up to 4 visits
  Prediction models of postprandial plasma glucose in relation to the macronutrient content of predefined meals as assessed by plasma and/or ISF concentrations of amino acids, glucose, and/or triglycerides

SECONDARY OUTCOMES:
Amino acid metabolism | Up to 14 hours per study visit, up to 4 visits
  Prediction models of postprandial plasma amino acid patterns in relation to the macronutrient content of predefined meals as assessed by plasma and/or ISF concentrations of amino acids and/or glucose

CONTACTS AND LOCATIONS:
Overall Officials: Nicolaas Deutz, MD, PhD, Principal Investigator — Texas A&M University; Michael McShane, PhD, Principal Investigator — Texas A&M University
Locations (1):
- Center for Translational Research in Aging & Longevity, College Station, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Data may be shared upon request based on methods/proposals approved by both parties' institutional review committees. Individual participant data that underlie the results of the trial may be shared after de-identification (text, tables, figures, and appendices). Additional documents available per request including: study protocol, statistical analysis plan, and informed consent.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: up to 6 years beyond the completion of the trial
Access Criteria: Contact PI - Dr. Michael McShane (mcshane@tamu.edu)

DOCUMENTS (2):
  • Study Protocol (2024-04-10): https://cdn.clinicaltrials.gov/large-docs/81/NCT06582381/Prot_000.pdf
  • Informed Consent Form (2024-02-23): https://cdn.clinicaltrials.gov/large-docs/81/NCT06582381/ICF_001.pdf